CLINICAL TRIAL: NCT02300064
Title: Mechanisms of Adaptation to Exercise in Health and Chronic Obstructive Pulmonary Disease (COPD); Oxidative Stress Links Aging, Activity and Mobility
Brief Title: Exercise in Health and Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Russell Richardson, Ph.D., University of Utah
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 32404
Record Dates: First submitted 2014-11-14; First posted 2014-11-24 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Exercise Test; Magnetic Resonance Spectroscopy; Antioxidants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Healthy volunteers (Experimental): Healthy volunteers will undergo one or more exercise interventions: knee-extensor exercise test; exercise test with restricting/releasing blood flow; exercise test with variable oxygen concentration and MRI; or exercise test with oral antioxidant or placebo cocktail.
  Interventions: Other: Knee-extensor exercise test; Other: Exercise test with restricting/releasing blood flow; Other: Exercise test with variable oxygen concentration and MRI; Other: Exercise test with oral antioxidant or placebo cocktail
- COPD patients (Experimental): Patients with Chronic Obstructive Pulmonary Disease (COPD) will undergo one or more exercise interventions: knee-extensor exercise test; exercise test with restricting/releasing blood flow; exercise test with variable oxygen concentration and MRI; or exercise test with oral antioxidant or placebo cocktail.
  Interventions: Other: Knee-extensor exercise test; Other: Exercise test with restricting/releasing blood flow; Other: Exercise test with variable oxygen concentration and MRI; Other: Exercise test with oral antioxidant or placebo cocktail

INTERVENTIONS:
Other: Knee-extensor exercise test — Steady-state, single leg knee-extensor exercise at 20 Watts for 10 minutes
Other: Exercise test with restricting/releasing blood flow — 10 minute submaximal (20 Watts) single leg knee-extensor exercise with blood flow clamped 10-15% lower by arterial infustion of phenylephrine; 10 minute passive single leg knee-extensor exercise with blood flow matched to the 20 Watt work rate level by arterial adenosine infusion; 10 minute seated rest with blood flow matched to the 20 Watt work rate level by adenosine infusion. Each test separated by at least 30 minutes rest.
Other: Exercise test with variable oxygen concentration and MRI — Two bouts of single leg knee-extensor exercise to maximal effort breathing regular air (21% oxygen) or 100% oxygen through a mouthpiece, with a 90 minute rest period between each bout. The same experiment performed again on a separate day in an magnetic resonance imaging (MRI) machine
Other: Exercise test with oral antioxidant or placebo cocktail — Antioxidants (Vitamin E - 400 international units, Vitamin C - 1000 milligrams and Alpha lipoic acid - 600 milligrams) or matching placebo capsules administered orally followed by femoral nerve stimulation and single leg knee-extensor exercise for 30 minutes at 50% maximum effort

SUMMARY:
The purpose of this study is to find out more about the effects of chronic obstructive pulmonary disease (COPD) on the function of blood vessels, the heart, and muscle at rest and during exercise.

DETAILED DESCRIPTION:
Oxidative stress, defined as an imbalance between pro and antioxidant molecular species in favor of the former, has recently been recognized as a potential mechanism in the peripheral muscle dysfunction associated with COPD. a series of studies are proposed to better understand the role and source of oxidative stress in the skeletal muscle of patients with COPD. Specifically, three main aims will address the following questions regarding COPD, skeletal muscle, and oxidative stress: where is oxidative stress most prevalent, why does oxidative stress occur, and what are the consequences of oxidative stress in COPD? the overall hypothesis to be tested is that COPD results in a shift toward greater intramuscular oxidative stress and this is, at least in part, responsible for the diminished mechanical efficiency and greater peripheral muscle fatiguability during muscular work often associated with this disease. The vascular consequence of this augmented free radical load is altered vascular function and a disruption of the local matching of perfusion and metabolism in skeletal muscle during exercise. These crucial changes result in a cascade of factors such as local hypoxia and elevated vascular shear stress, entering a vicious cycle that leads to the generation of more free radicals, especially during physical work. It is proposed that this imbalance between pro and antioxidant potential, toward oxidative stress, plays a significant role in the attenuated exercise capacity and reduced muscle fatigue resistance associated with COPD.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Obstructive Pulmonary Disease (COPD) patients (over 18 years old) and
* age-matched healthy controls (over 18 years old)

Exclusion Criteria:

* Severe Chronic Obstructive Pulmonary Disease (volume exhaled at the end of the first section of forced expiration is predicted to be under 30 percent),
* Severe Heart Failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2009-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change in Free Radical Concentration in Muscle Tissue Following Exercise | Baseline to two hours

SECONDARY OUTCOMES:
Change in Free Radical Concentration in Muscle Venous Outflow following Exercise | Baseline to two hours

CONTACTS AND LOCATIONS:
Overall Officials: Russell Richardson, Ph.D., Principal Investigator — US Department of Veterans Affairs
Locations (1):
- Veterans Affairs Salt Lake City Heath Care System, Salt Lake City, Utah, United States